CLINICAL TRIAL: NCT00618982
Title: A Phase II, Multi-centre, Open-label Study to Assess the Efficacy, Safety, Tolerability and Pharmacokinetics of Intrapatient Dose Escalation of Sorafenib as First Line Treatment for Metastatic Renal Cell Carcinoma.
Brief Title: Sorafenib Dose Escalation in Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12913; 2007-004875-21 (EudraCT Number)
Record Dates: First submitted 2008-02-08; First posted 2008-02-20 (Estimated); Results first posted 2010-05-27 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-11

CONDITIONS: Carcinoma, Renal Cell
Keywords: Kidney cancer,; Sorafenib,; Dose escalation,; No previous treatment
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib (Nexavar, BAY43-9006) (Experimental): Intrapatient dose escalation of sorafenib from 400 mg orally twice daily (bid) for the first cycle, 600 mg bid for the second cycle and 800 mg bid until disease progression, unacceptable toxicity or withdrawal of consent. Dose reductions due to toxicities were allowed.
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — The initial dose of sorafenib will be 400 mg bid administered orally, on a continuous basis. A treatment cycle is considered to be 28 days. Intrapatient dose escalation will occur according to the following schedule, providing no grade 3 or 4 toxicities are observed (except for alopecia, nausea and vomiting); Day 1-28 400 mg bid, Day 29-56 600 mg bid, Day 57 onwards 800 mg bid. Subjects will continue on treatment until progression, unacceptable toxicity, subject withdraws consent or the decision is taken to stop the study following the analysis of response rates.

SUMMARY:
Sorafenib is a new drug, which is approved under the brand name Nexavar for the treatment of advanced kidney cancer. It is also currently being tested in various other cancers. Sorafenib works by stopping the development of new cancer cells and new blood vessels. By stopping the growth of new blood vessels around a tumor, it is believed that sorafenib prevents the growth of kidney cancer tumors.

This is an "open-label" study which means that the patient, the doctor and Bayer Healthcare will know what tablets the patient is taking. All patients in this study will receive sorafenib tablets. Sorafenib is taken orally as a tablet (two tablets are taken twice a day). Treatment with sorafenib will continue until the patient's tumor grows larger or spreads further or if the patient has intolerable side effects. The dose of sorafenib that the patient will receive in the study will increase at certain points during the patient's treatment, as long as the patient is not experiencing side effects and the patient's tumor has not grown.

DETAILED DESCRIPTION:
Issues on Outcome Measure "Safety and tolerability" will be addressed in the Adverse Events section.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Metastatic clear cell RCC (renal cell carcinoma)
* Subjects with at least one uni-dimensional measurable lesion.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Memorial Sloan Kettering Cancer Center (MSKCC) good or intermediate category
* Life expectancy of at least 12 weeks.
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to treatment
* Signed informed consent must be obtained prior to any study specific procedures.
* Subjects must have received no prior systemic anticancer therapy for the treatment of their renal cell carcinoma
* Prior total nephrectomy

Exclusion Criteria:

* History of cardiac disease
* History of human immunodeficiency virus (HIV) infection or chronic hepatitis B or C
* Active clinically serious infections (> grade 2 National Cancer Institute-Common Terminology Criteria for Adverse Events [NCI-CTCAE] version 3.0)
* Symptomatic metastatic brain or meningeal tumors unless the subject is > 6 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable with respect to the tumor at the time of study entry.
* Subjects with evidence or history of bleeding diathesis
* Deep vein thrombosis and/or pulmonary embolus within 12 months of the start of treatment.
* Delayed healing of wounds, ulcers or bone fractures
* Subjects with pre-existing thyroid abnormality whose thyroid function cannot be maintained within the normal range by medication
* Subjects undergoing renal dialysis
* Pregnant or breast-feeding subjects. Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and three months after the completion of trial.
* Prior adjuvant sorafenib is excluded.
* Radiotherapy during study or within 3 weeks of start of study drug
* Major surgery within 4 weeks of start of study
* Investigational drug therapy outside of this trial during or within 4 weeks of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2008-02; Primary Completion 2009-04 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (21):
- France (6):
  - Bordeaux
  - La Roche-sur-Yon
  - Marseille
  - Nantes
  - Paris
  - Tours
- Germany (5):
  - Tübingen, Baden-Wurttemberg
  - Marburg, Hesse
  - Hanover, Lower Saxony
  - Mainz, Rhineland-Palatinate
  - Jena, Thuringia
- Italy (3):
  - Aviano, Pordenone
  - Milan
  - Pavia
- Poland (3):
  - Olsztyn
  - Warsaw
  - Wroclaw
- United Kingdom (4):
  - London, London
  - Greater Manchester, Manchester
  - Cardiff, South Glamorgan
  - Glasgow

REFERENCES:
- See also: Click here and search for Bayer product information provided by EMA — http://www.clinicaltrialsregister.eu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 04 Feb to 05 Nov 2008 at 19 centers in 5 countries (Germany, France, United Kingdom, Italy and Poland).
Pre-assignment Details: Of the 89 subjects enrolled, 83 were treated with the study drug. Safety population = 83 subjects who took at least one dose of study drug and had any data after baseline. Intent to treat population = 67 subjects treated with the study drug who had at least one efficacy evaluation after baseline.
Period: Overall Study
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Started | 83
Completed | 33
Not Completed | 50
Not completed — Adverse Event | 23
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1
Not completed — ongoing, still treated with study med. | 25

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 83
Age, Continuous [Median (Full Range); unit: years] | 61 [33 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 54
ECOG (Eastern Cooperative Oncology Group) Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is a scale that measures how cancer affects the daily life of a patient on an ordinal scale from grade 0 (best) to grade 5 (worst). Status 0 = fully active; Status 1 = restricted strenuous activity, ambulatory and able to carry out work of a light or sedentary nature
  participants
    0 | 49
    1 | 34
Stage at study entry [Number; unit: participants] — Categorized information on tumor size, lymph node involvement and metastases. Stages I-IV. The higher the stage, the more advanced cancer.
  participants
    Stage III | 1
    Stage IV | 82

OUTCOME MEASURES:

1. Primary Outcome: Best Response - mITT (Modified Intent-to-treat) Population
Description: Best Response (Response Rate) of a subject was defined as the proportion of patients with confirmed Complete Response (CR) or Partial Response (PR) as their best response observed (by independent central assessment) during trial period assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST version 1.0) criteria. Confirmed CR was defined as disappearance of tumor and PR was defined as a decrease of at least 30% in the sum of tumor lesion sizes.
Time Frame: Radiological assessments were performed every 8 weeks (2 cycles) from start of the treatment. After completion of 6 cycles of treatment at the highest tolerated dose level, assessments were performed every 12 weeks for up to 34 months.
Population: The population for the analysis of primary efficacy variable was the modified intent-to-treat (mITT) population defined as the patients treated for at least 6 months with 4 months at their highest tolerated dose.
Measure: Number; unit: Participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 18
Participants | 8 [21.5 to 69.2]

2. Primary Outcome: Tumor Response - ITT (Intent to Treat) Population
Description: Tumor Response of a subject was defined as the best tumor response observed (by independent central assessment) during trial period assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST version 1.0) criteria. Confirmed Complete Response (CR) was defined as disappearance of tumor, Partial Response (PR) was defined as a decrease of at least 30% in the sum of target lesions, Stable Disease (SD) was defined as steady state of disease, and Progressive Disease (PD) was defined as at least a 20% increase in the sum of measured lesions or appearance of new lesions.
Time Frame: as for outcome 1
Population: The population for the efficacy analysis was the intent-to-treat (ITT) population defined as all patients who received at least one dose of study medication with at least one valid tumor assessment post-baseline.
Measure: Number; unit: participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 67
participants
  Complete Response (CR) | 0
  Partial Response (PR) | 12
  Stable Disease (SD) | 46
  Progressive Disease (PD) | 9

3. Secondary Outcome: Pharmacokinetics (PK) Analysis - Area Under the Drug Concentration-time Curve From Time Zero to 10 Hours Postdose (AUC(0-10),ss)
Description: AUC(0-10),ss was defined as an area under the plasma concentration versus time curve from time zero to 10 hours post-dose. Parameter was calculated for sorafenib and M2, an active metabolite of sorafenib.
Time Frame: Blood samples were collected at screening (blank) and on day 28 of the first cycle completed at each dose level. Samples were drawn at the following time points in relation to morning dose of sorafenib: pre-dose, 2, 4, 6, 8 and 10 hours post-dose.
Population: PK Analysis Population. 40 participants in the 400 mg bid group that had an AUC(0-10)ss calculated; 30 participants in the 600 mg bid group that had an AUC(0-10)ss calculated; 26 participants and 27 participants in the 800 mg bid group that had an AUC(0-10)ss calculated, for sorafenib and M2 parameter respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*h/L
Groups:
- Sorafenib (Nexavar, BAY43-9006)_400 mg: Participants received 400 mg orally twice daily (bid)
- Sorafenib (Nexavar, BAY43-9006)_600 mg: Participants received 600 mg orally twice daily (bid)
- Sorafenib (Nexavar, BAY43-9006)_800 mg: Participants received 800 mg orally twice daily (bid)
Arm/Group | Sorafenib (Nexavar, BAY43-9006)_400 mg | Sorafenib (Nexavar, BAY43-9006)_600 mg | Sorafenib (Nexavar, BAY43-9006)_800 mg
Number analyzed (Participants) | 40 | 30 | 26
mg*h/L
  Sorafenib (N=40, 30, 26) | 50.0 (39.2) | 51.2 (43.7) | 43.8 (47.8)
  M2 (BAY67-3472) (N=40, 30, 27) | 8.80 (74.3) | 10.4 (82.1) | 8.23 (87.2)

4. Secondary Outcome: Pharmacokinetics (PK) Analysis - Area Under the Drug Concentration-time Curve From Time Zero to 12 Hours Postdose (AUC(0-12),ss)
Description: AUC(0-12),ss was defined as an area under the plasma concentration versus time curve from time zero to 12 hours post-dose. Parameter was calculated for sorafenib and M2, an active metabolite of sorafenib.
Time Frame: Blood samples were collected at screening (blank) and on day 28 of the first cycle completed at each dose level. Samples were drawn at the following time points in relation to morning dose of sorafenib: pre-dose, 2, 4, 6, 8, 10 and 12 hours post-dose.
Population: PK Analysis Population. 32 participants in the 400 mg bid group that had an AUC(0-12)ss calculated; 23 participants in the 600 mg bid group that had an AUC(0-12)ss calculated; 19 participants and 20 participants in the 800 mg bid group that had an AUC(0-12)ss calculated, for sorafenib and M2 parameter respectively.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*h/L
Arm/Group | Sorafenib (Nexavar, BAY43-9006)_400 mg | Sorafenib (Nexavar, BAY43-9006)_600 mg | Sorafenib (Nexavar, BAY43-9006)_800 mg
Number analyzed (Participants) | 32 | 23 | 19
mg*h/L
  Sorafenib (N=32, 23, 19) | 57.2 (39.1) | 57.6 (46.1) | 47.0 (51.9)
  M2 (BAY67-3472) (N=32, 23, 20) | 9.58 (78.2) | 11.2 (75.9) | 8.41 (94.6)

5. Secondary Outcome: Pharmacokinetics (PK) Analysis - Maximum Observed Concentration in Plasma (Cmax)
Description: Cmax was defined as a maximum plasma concentration at steady-state. Parameter was calculated for sorafenib and M2, an active metabolite of sorafenib.
Time Frame: as for outcome 4
Population: PK Analysis Population. 40 participants in the 400 mg bid group that had Cmax calculated; 31 participants in the 600 mg bid group that had Cmax calculated; 28 participants in the 800 mg bid group that had Cmax calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Sorafenib (Nexavar, BAY43-9006)_400 mg | Sorafenib (Nexavar, BAY43-9006)_600 mg | Sorafenib (Nexavar, BAY43-9006)_800 mg
Number analyzed (Participants) | 40 | 31 | 28
mg/L
  Sorafenib | 7.53 (38.0) | 7.62 (39.3) | 6.64 (42.1)
  M2 (BAY67-3472) | 1.31 (80.8) | 1.51 (81.4) | 1.30 (88.5)

6. Secondary Outcome: Pharmacokinetics (PK) Analysis - Time to Maximum Concentration (Tmax)
Description: Tmax was defined as a time to maximum concentration at steady-state. Parameter was calculated for sorafenib and M2, an active metabolite of sorafenib.
Time Frame: as for outcome 4
Population: PK Analysis Population. 40 participants in the 400 mg bid group that had Tmax calculated; 31 participants in the 600 mg bid group that had Tmax calculated; 28 participants in the 800 mg bid group that had Tmax calculated.
Measure: Median (Full Range); unit: hours
Arm/Group | Sorafenib (Nexavar, BAY43-9006)_400 mg | Sorafenib (Nexavar, BAY43-9006)_600 mg | Sorafenib (Nexavar, BAY43-9006)_800 mg
Number analyzed (Participants) | 40 | 31 | 28
hours
  Sorafenib | 2 [0.00 to 12.0] | 2 [0.00 to 12.0] | 2 [0.00 to 12.0]
  M2 (BAY67-3472) | 2 [0.00 to 10.3] | 2 [0.00 to 12.0] | 1 [0.00 to 12.0]

7. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) was defined as the time from start of study medication to the first documented disease progression per RECIST (by independent radiological assessment) or clinical progression as per investigator assessment or death due to any cause whichever occurred first. For patients who had not recurred or died at the time of analysis, PFS was censored at their last date of evaluable scan.
Time Frame: as for outcome 1
Population: Intent-to-treat (ITT).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 67
months | 7.4 [6.0 to 11.7]

8. Secondary Outcome: Time to Progression (TTP)
Description: Time to progression (TTP) was defined as the time from start of study medication to the first documented disease progression per RECIST (by independent radiological assessment) or clinical progression as per investigator assessment whichever occurred first. For patients who had not progressed at the time of analysis or died before progression, TTP was censored at their last date of evaluable scan.
Time Frame: as for outcome 1
Population: Intent-to treat (ITT).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 67
months | 7.4 [6.0 to 11.7]

9. Other Pre Specified Outcome: Tumor Response - mITT Population
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 18
Participants
  Complete response (CR) | 0
  Partial response (PR) | 8
  Stable disease (SD) | 10
  Progressive disease (PD) | 0

10. Other Pre Specified Outcome: Disease Control - mITT Population
Description: Disease Control (DC) of a subject was defined as the proportion of patients with confirmed Complete Response (CR), Partial Response (PR) or Stable Disease (SD) as their best response observed (by independent central assessment) during trial period assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST version 1.0) criteria. Confirmed CR was defined as disappearance of tumor, PR was defined as a decrease of at least 30% in the sum of tumor lesion sizes, and SD was defined as steady state of disease.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 18
Participants | 18 [81.5 to 100]

ADVERSE EVENTS:
Description: Abbreviations used in the Adverse Events section: Gastrointestinal (GI), Not Otherwise Specified (NOS), Absolute Neutrophil Count (ANC), Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Gamma glutamyl transpeptidase (GGT)
Groups:
- Sorafenib (Nexavar, BAY43-9006): Intrapatient dose escalation of sorafenib from 400 mg orally twice daily (bid) for the first cycle,600 mg bid for the second cycle and 800 mg bid until disease progression, unacceptable toxicity or withdrawal of consent. Dose reductions due to toxicities were allowed.
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Serious Adverse Events (participants affected / at risk) | 45/83
Other Adverse Events (participants affected / at risk) | 80/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) (N=83)
Hemoglobin (Blood and lymphatic system disorders) | 1
Cardiac arrhythmia - Other (Cardiac disorders) | 2
Cardiac general - Other (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
GI - Other (Gastrointestinal disorders) | 3
Constitutional symptoms - Other (General disorders) | 1
Fatigue (General disorders) | 3
Fever (General disorders) | 1
Pain, Abdomen NOS (General disorders) | 1
Pain, Back (General disorders) | 2
Pain, Bone (General disorders) | 1
Pain, Breast (General disorders) | 1
Pain, Chest/Thorax NOS (General disorders) | 1
Pain, Joint (General disorders) | 1
Pain, Other (General disorders) | 1
Pain, Stomach (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Hepatobiliary - Other (Hepatobiliary disorders) | 2
Allergic reaction (Immune system disorders) | 1
Infection (Documented clinically), Kidney (Infections and infestations) | 1
Infection (Documented clinically), Lung (Pneumonia) (Infections and infestations) | 2
Infection with normal ANC, Abdomen NOS (Infections and infestations) | 1
Infection with normal ANC, Anal/perianal (Infections and infestations) | 1
Infection with normal ANC, Sinus (Infections and infestations) | 1
Intraop injury - Other (Injury, poisoning and procedural complications) | 3
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal - Other (Musculoskeletal and connective tissue disorders) | 2
Secondary malignancy (possibly related to cancer treatment) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Confusion (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Neurology - Other (Nervous system disorders) | 1
Neuropathy: motor (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Airway obstruction, Bronchus (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Dermatology - Other (Skin and subcutaneous tissue disorders) | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3
Thrombosis/Thrombus/Embolism (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) (N=83)
Edema: Limb (Blood and lymphatic system disorders) | 7
Hemoglobin (Blood and lymphatic system disorders) | 12
Neutrophils (Blood and lymphatic system disorders) | 3
Platelets (Blood and lymphatic system disorders) | 7
Hypertension (Cardiac disorders) | 40
Hypotension (Cardiac disorders) | 3
Hyperthyroidism (Endocrine disorders) | 3
Hypothyroidism (Endocrine disorders) | 12
Dry eye (Eye disorders) | 3
Ocular - Other (Eye disorders) | 3
Anorexia (Gastrointestinal disorders) | 21
Colitis (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 53
Dry mouth (Gastrointestinal disorders) | 3
GI - Other (Gastrointestinal disorders) | 13
Gastritis (Gastrointestinal disorders) | 3
Heartburn (Gastrointestinal disorders) | 8
Hemorrhoids (Gastrointestinal disorders) | 3
Mucositis (clinical exam), Oral cavity (Gastrointestinal disorders) | 6
Mucositis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 28
Nausea (Gastrointestinal disorders) | 22
Taste Alteration (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 16
Constitutional symptoms - Other (General disorders) | 15
Fatigue (General disorders) | 45
Fever (General disorders) | 14
Flu-like syndrome (General disorders) | 6
Insomnia (General disorders) | 4
Pain, Abdomen NOS (General disorders) | 10
Pain, Back (General disorders) | 8
Pain, Bone (General disorders) | 4
Pain, Breast (General disorders) | 3
Pain, Chest wall (General disorders) | 3
Pain, Chest/Thorax NOS (General disorders) | 5
Pain, Dental/Teeth/peridontal (General disorders) | 4
Pain, Extremity - limb (General disorders) | 8
Pain, Head/Headache (General disorders) | 7
Pain, Joint (General disorders) | 6
Pain, Muscle (General disorders) | 5
Pain, Other (General disorders) | 6
Pain, Stomach (General disorders) | 5
Weight loss (General disorders) | 14
Allergy - Other (Immune system disorders) | 3
Infection (Documented clinically), Bladder (urinary) (Infections and infestations) | 6
Infection (Documented clinically), Skin (Cellulitis) (Infections and infestations) | 3
Infection (Documented clinically), Urinary tract NOS (Infections and infestations) | 3
Infection - Other (Infections and infestations) | 3
ALT (Metabolism and nutrition disorders) | 7
AST (Metabolism and nutrition disorders) | 6
Amylase (Metabolism and nutrition disorders) | 5
Creatinine (Metabolism and nutrition disorders) | 4
GGT (Metabolism and nutrition disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 5
Hyperuricemia (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 7
Hypokalemia (Metabolism and nutrition disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 16
Lipase (Metabolism and nutrition disorders) | 16
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 7
Musculoskeletal - Other (Musculoskeletal and connective tissue disorders) | 10
Dizziness (Nervous system disorders) | 4
Mood Alteration, Anxiety (Nervous system disorders) | 4
Mood alteration, Depression (Nervous system disorders) | 6
Neurology - Other (Nervous system disorders) | 4
Neuropathy: sensory (Nervous system disorders) | 12
Cystitis (Renal and urinary disorders) | 3
Renal - Other (Renal and urinary disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Dyspnea (Shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 15
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 3
Voice changes (Respiratory, thoracic and mediastinal disorders) | 11
Alopecia (Skin and subcutaneous tissue disorders) | 36
Dermatology - Other (Skin and subcutaneous tissue disorders) | 19
Dry skin (Skin and subcutaneous tissue disorders) | 23
Erythema multiforme (Skin and subcutaneous tissue disorders) | 6
Flushing (Skin and subcutaneous tissue disorders) | 5
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 54
Nail changes (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 15
Rash/desquamation (Skin and subcutaneous tissue disorders) | 46
Hemorrhage pulmonary, Nose (Vascular disorders) | 3
Hemorrhage, GI, Oral cavity (Vascular disorders) | 4
Thrombosis/Thrombus/Embolism (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator (PI) can publish results following completion of study. The PI must discuss a publication with Bayer prior to release&obtain written consent to proceed. The Investigator must send a draft to Bayer at least 30d in advance of submission to obtain approval. Any submission to Bayer will be reviewed w/o unreasonable delay&approval not be withheld unreasonably. In difference of opinion publication will be discussed.